CLINICAL TRIAL: NCT04997252
Title: An Evaluation of the Efficacy and Safety of Apalutamide as Neoadjuvant Endocrine Therapy in High-Risk and Oligometastatic Prostate Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Principal Investigator, Binshen Chen, associate chief physician, Zhujiang Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Chen-001
Record Dates: First submitted 2021-07-29; First posted 2021-08-09 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: High-Risk and Oligometastatic Prostate Cancer
MeSH Terms: interventions — apalutamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- high-risk and oligometastatic prostate cance (Experimental): Neoadjuvant therapy with apalutamide in combination with luteinizing hormone-releasing hormone analogues
  Interventions: Drug: Apalutamide

INTERVENTIONS:
Drug: Apalutamide — apalutamide as neoadjuvant therapy

SUMMARY:
The neoadjuvant therapy with apalutamide can significantly improve the prognosis of patients with high-risk and oligometastatic prostate cancer, lower the rate of positive margins, reduce recurrence, and show high safety.

ELIGIBILITY:
Inclusion Criteria:

1. Adult males aged above 18 years old, no healthy volunteers included;
2. Prostate cancer confirmed by pathological findings;
3. High risk based on risk assessment, or laboratory tests suggestive of oligometastasis;
4. Agreement to undergo laparoscopic radical prostatectomy + pelvic lymphadenectomy;
5. ECOG score of 0 - 1
6. Agreement to undergo preoperative and postoperative endocrine therapy;
7. Voluntary signing of an ICF for the clinical trial

Exclusion Criteria:

1. Any other tumor disease requiring treatment;
2. Any organ metastasis confirmed by imaging, such as liver and brain metastases, or the possibility of paralysis due to spinal cord metastasis;
3. A history of epilepsy or any condition that may lead to seizures;
4. Severe liver or kidney dysfunction, severe cardiovascular or cerebrovascular diseases, and systemic immune system diseases.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
rPFS | Change from Baseline at preoperative 1, 2, and 3 months and postoperative 1, 3, 6, 9, 12, 18, and 24 months.
  radiographic progression-free survival

SECONDARY OUTCOMES:
pCR | preoperative 1, 2, and 3 months and postoperative 1, 3, 6, 9, 12, 18, and 24 months.
  pathological complete response
PFS | preoperative 1, 2, and 3 months and postoperative 1, 3, 6, 9, 12, 18, and 24 months.
  positive margin rate; progression-free survival
PSA response rate: | preoperative 1, 2, and 3 months and postoperative 1, 3, 6, 9, 12, 18, and 24 months.
  more than 50% decrease from baseline
TTPP | preoperative 1, 2, and 3 months and postoperative 1, 3, 6, 9, 12, 18, and 24 months.
  time to PSA progression
time to BCR after surgery | preoperative 1, 2, and 3 months and postoperative 1, 3, 6, 9, 12, 18, and 24 months.
pathological stage | preoperative 1, 2, and 3 months and postoperative 1, 3, 6, 9, 12, 18, and 24 months.

CONTACTS AND LOCATIONS:
Locations (1):
- zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong, China